CLINICAL TRIAL: NCT00087165
Title: A Phase II Study of GTI-2040 in Combination With Docetaxel and Prednisone in Hormone-Refractory Prostate Cancer
Brief Title: GTI-2040, Docetaxel, and Prednisone in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: PMH-PHL-024; CDR0000372951 (Registry Identifier: PDQ (Physician Data Query)); NCI-6102
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — GTI2040; Docetaxel; Prednisone

INTERVENTIONS:
Biological: GTI-2040
Drug: docetaxel
Drug: prednisone

SUMMARY:
RATIONALE: GTI-2040 may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. GTI-2040 may help docetaxel kill more tumor cells by making them more sensitive to the drug.

PURPOSE: This phase II trial is studying how well giving GTI-2040 together with docetaxel and prednisone works in treating patients with prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of GTI-2040, docetaxel, and prednisone, in terms of prostate-specific antigen (PSA) response rate, in patients with hormone-refractory prostate cancer.

Secondary

* Determine objective tumor response in patients treated with this regimen.
* Determine the median time to progression in patients treated with this regimen.
* Determine the safety and tolerability of this regimen in these patients.
* Determine the median duration of PSA response in patients treated with this regimen.
* Correlate baseline and post-treatment levels of ribonucleotide reductase activity in tumor biopsies and peripheral blood mononuclear cells and tumoral expression of c-myc, R2 subunit protein, and markers of cellular proliferation and apoptosis with clinical outcomes in patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study.

Patients receive GTI-2040 IV continuously on days 1-14, docetaxel IV on day 3 of course 1 and on day 1 of subsequent courses, and oral prednisone twice daily on days 1-21. Treatment repeats every 21 days for up to 10 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 18-46 patients will be accrued for this study within 3.6-9.5 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Histologically or cytologically confirmed adenocarcinoma of the prostate
  * Metastatic carcinoma of presumptive prostate origin

    * Bony metastases AND a serum prostate-specific antigen (PSA) level > 20 ng/mL
* Disease progression after prior hormonal therapy as defined by rising PSA levels

  * At least 2 consecutive rises in PSA over a reference value, with measurements taken at least 7 days apart
  * Prior hormonal therapy must include either medical (luteinizing hormone-releasing hormone [LHRH] agonist) OR surgical (orchiectomy) castration

    * Patients who received prior LHRH agonist must continue or re-start such therapy
* Castrate levels of testosterone < 50 ng/dL
* PSA ≥ 20 ng/mL
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* WBC ≥ 3,000/mm^3

Hepatic

* AST and ALT ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin normal
* PTT ≤ 1.25 times upper limit of control
* INR ≤ 1.3

Renal

* Creatinine ≤ 1.5 times ULN OR
* Creatinine clearance ≥ 50 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Fertile patients must use effective contraception
* No symptomatic peripheral neuropathy ≥ grade 2
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to GTI-2040 or other study agents
* No concurrent uncontrolled illness
* No active or ongoing infection
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent prophylactic filgrastim (G-CSF) or epoetin alfa

Chemotherapy

* No prior chemotherapy except monotherapy with oral estramustine
* At least 4 weeks since prior estramustine and recovered

Endocrine therapy

* See Disease Characteristics
* At least 6 weeks since prior bicalutamide*
* At least 4 weeks since prior flutamide, nilutamide, or cyproterone*
* Concurrent steroids allowed NOTE: *Patients must have evidence of disease progression despite cessation of antiandrogen therapy

Radiotherapy

* At least 4 weeks since prior radiotherapy
* No prior radiotherapy to > 25% of bone marrow
* No prior isotope therapy

Surgery

* See Disease Characteristics

Other

* No concurrent prophylactic antibiotics
* No concurrent anticoagulants

  * Concurrent low-dose warfarin for prophylaxis of central line thrombosis allowed
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents or therapies

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2006-09 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
PSA response rate

SECONDARY OUTCOMES:
Median survival
1-year survival
Response rate and duration

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm J. Moore, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (5):
- Canada (5):
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Result] Sridhar SS, Canil CM, Chi KN, Hotte SJ, Ernst S, Wang L, Chen EX, Juhasz A, Yen Y, Murray P, Zwiebel JA, Moore MJ. A phase II study of the antisense oligonucleotide GTI-2040 plus docetaxel and prednisone as first-line treatment in castration-resistant prostate cancer. Cancer Chemother Pharmacol. 2011 Apr;67(4):927-33. doi: 10.1007/s00280-010-1389-7. Epub 2010 Jul 3. PMID 20602233